CLINICAL TRIAL: NCT04917809
Title: A Phase 2 "Window of Opportunity" Trial of Targeted Therapy With Erdafitinib in Patients With Recurrent FGFR3-Altered Non-Muscle Invasive Bladder Cancer
Brief Title: A Study of Oral Erdafitinib in People With Recurrent Non-Invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-166
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Bladder Cancer; Recurrent Bladder Cancer; FGFR3 Gene Mutation
Keywords: Non-Muscle Invasive Bladder Cancer; NMIBC; Erdafitinib; FGFR3; 21-166; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with FGFR3-mutant or -fusion noninvasive bladder tumors (Experimental): 25 participants with FGFR3-mutant or -fusion noninvasive bladder tumors will be accrued.
  Interventions: Drug: Erdafitinib

INTERVENTIONS:
Drug: Erdafitinib — Participants will receive erdafitinib at a dose of 6 mg orally once daily for the first 14 days (±3 days). Serum phosphate levels will be assessed on day 14 (±3 days) and the dose of erdafitinib may be lowered based on the serum phosphate level. Treatment with erdafitinib at a dose of 6 mg orally once daily, or at a lower dose level for another 14 days (±3 days) until the day of their standard-of-care TURBT/biopsy. Standard-of-care TURBT/biopsy will be performed after approximately 28 days (±5 days) from the start of treatment with erdafitinib, and biologic and pathologic tumor response will be assessed. All participants will then be followed up for recurrence or progression in accordance with the standard of care.

SUMMARY:
The purpose of this study is to assess the effectiveness of erdafitinib in people with non-muscle invasive bladder cancer (NMIBC) that has come back after standard treatment, such as Bacillus Calmette-Guerin (BCG) or chemotherapy instilled into the bladder. Participants in this study will have bladder cancer with a mutation in the FGFR3 gene. FGFR3 mutations are the most common genetic alteration in NMIBC and is present in the majority of recurrent NMIBC tumors. Genetic testing of the participant's prior or recurrent NMIBC tumor will be performed to confirm it has an FGFR3 gene mutation. Erdafitinib is a pill given orally (by mouth) that blocks the protein made by this altered gene, which may stop cancer cells from growing. Erdafitinib is already used as an approved treatment for metastatic bladder cancer. Researchers are doing this study to determine whether erdafitinib is an effective treatment for FGFR3-altered non-muscle invasive bladder cancer in the time period between when a recurrent tumor is identified and a TURBT (transurethral resection of a bladder tumor) or biopsy procedure is performed to remove it.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have NMIBC that has come back after prior treatment (instillations of BCG or chemotherapy into the bladder).
* Genetic testing of the participant's prior or recurrent NMIBC tumor will be performed to confirm the presence of an FGFR3 mutation
* Patients must be able to walk and do routine activities for more than half of their normal waking hours.
* This study is for people age 18 and older.
* Willing and able to provide written informed consent for the trial.
* Documentation on MSK-IMPACT of an oncogenic FGFR3 mutation (R248C, S249C, G370C, Y373C, etc.) or FGFR3 gene fusion with compelling clinical or biologic evidence in the OncoKB Precision Oncology Knowledge Base (https://oncokb.org/) from either archival NMIBC tumor tissue or recent TURBT/biopsy specimen of current tumor tissue.
* Any recurrence of noninvasive-appearing papillary tumor(s) (clinical Ta disease) after at least 1 previous course of intravesical therapy with either:

  * (1) a history of a high-grade Ta tumor -OR-
  * (2) a history of low-grade T1 tumor -OR-
  * (3) low-grade Ta tumor with the new recurrent tumor demonstrating at least 1 additional "unfavorable" risk factor for future recurrence:
* Multiple tumors
* Tumor size ≥3 cm
* Early recurrence ≤12 months from last treatment
* Frequent recurrences ≥1 per year

  ° Given the frequent shortages of BCG, a prior course of therapy with either BCG therapy or intravesical chemotherapy (mitomycin, gemcitabine, etc.) is acceptable. All prior treatments for NMIBC will recorded and described.
* Ages 18 or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Adequate bone marrow, liver, and renal function:

  ° Bone marrow function:
* Absolute neutrophil count (ANC) ≥1,000/mm3
* Platelet count ≥75,000/mm3
* Hemoglobin ≥8.0 g/dL

  ° Liver function:
* Total bilirubin ≤1.5 x ULN
* Alanine aminotransferase (ALT) ≤2.5 x ULN
* Aspartate aminotransferase (AST) ≤2.5x ULN

  ° Renal function:
* estimated glomerular filtration rate >30 mL/min/1.73m2 calculated using the modification of diet in renal disease equation or CKD-EPI formula
* Serum Phosphate level ≤ ULN prior to starting treatment
* Able to swallow pills
* Female subjects of childbearing potential should be on birth control, have male partners using a condom during intercourse, be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of the study therapy. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. While taking the study drug and for three months after the last dose of the study drug, sexually active males must use a condom during intercourse. They should not father a child during this period. Men who have undergone vasectomy are also required to use a condom during intercourse, to prevent delivery of the drug via seminal fluid.
* *Unless evaluated by a hematologist and decreased ANC is suspected to be caused by benign ethnic neutropenia (BEN) or DANC. Patient may proceed with treatment if deemed safe by a hematologist

Exclusion Criteria:

* Impaired decision-making capacity
* Pregnant (positive pregnancy test) or lactating.
* History of or currently being treated for muscle-invasive (i.e., stage T2 or higher) or metastatic urothelial cell carcinoma.
* Evidence of concurrent extravesical (i.e., urethra, ureter, or renal pelvis) urothelial cell carcinoma.
* Evidence of carcinoma in situ only disease (stage Tis) or concurrent carcinoma in situ.
* Patients who meet the definition BCG-unresponsive NMIBC as defined as:

  * HGT1 within 3 months after an induction BCG course (received ≥5 of 6 doses)
  * Persistent or recurrent high-grade NMIBC (Tis, Ta, T1) within 6 months of ≥5 of 6 doses of induction BCG therapy and ≥2 of 3 doses of maintenance BCG therapy
* History of or currently being treated for or scheduled to have radiation treatment for bladder cancer; prior radiation therapy for prostate cancer or another nonbladder cancer is allowed.
* Prior systemic chemotherapy, targeted therapy, or treatment with an investigational anticancer agent within 30 days or ≤5 half-lives of the agent (whichever is longer) before the first dose of erdafitinib.
* Prior immunotherapy within 30 days before the first dose of erdafitinib and/or has an ongoing grade ≥ 2 immunotherapy-related toxicity.
* Unstable angina, myocardial infarction within the preceding 3 months, or known New York Heart Association class II-IV congestive heart failure.
* Evidence of bleeding diathesis or coagulopathy.
* Cerebrovascular accident or transient ischemic attack within the preceding 3 months.
* Prior treatment with a selective FGFR inhibitor (including but not limited to AZD4547, BGJ398, BAY1163877, and LY2874455).
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of oral erdafitinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, and malabsorption syndrome).
* Current evidence of endocrine alterations of calcium/phosphate homeostasis (e.g., parathyroid disorders, history of parathyroidectomy, tumor lysis, and tumoral calcinosis).
* Use of medications that increase serum levels of phosphorus and/or calcium (e.g., calcium, phosphate, vitamin D, and parathyroid hormone). Patients on these medications can participate in the study if they are able to discontinue them while receiving treatment with erdafitinib.
* Use of medications that are known strong or moderate inhibitors or inducers of CYP3A4 or CYP2C9 (A comprehensive list is included in the Appendix: Drugs Classified as Strong or Moderate In Vivo Inhibitors and Inducers of CYP3A4/2C9 Enzymes). Patients on these medications can participate in the study if they are able to discontinue them prior to starting treatment with erdafitinib.
* Current evidence of corneal or retinal disorder/keratopathy, including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, and/or keratoconjunctivitis, confirmed by ophthalmologic examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 weeks after first study treatment
  The primary endpoint of this trial is the objective response rate at the time of TURBT/biopsy (defined as the proportion of patients achieving a complete or partial pathologic response by cytologic examination, cystoscopic examination, and biopsy) following treatment with erdafitinib. A complete response is defined as the absence of tumor on TURBT/biopsy, with a negative urinary cytologic result; a partial response is defined as a decrease of at least 50% in the size of the target tumor(s), on the basis of modified RECIST 1.1 criteria (RECIT-BLADDER).

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Pietzak, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org